CLINICAL TRIAL: NCT02415569
Title: Tailored Bowel Preparation According to Bristol Stool Form Scale: a Prospective, Randomized, Controlled, Investigator-blinded, Multicenter Study
Brief Title: Tailored Bowel Preparation According to Bristol Stool Form Scale
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Qianfoshan Hospital (Other); Binzhou People's Hospital (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2014SDU-QILU-G07
Record Dates: First submitted 2015-01-21; First posted 2015-04-14 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Bowel Cleansing Quality
Keywords: bowel cleansing; bisacodyl; polyethyleneglycol; colonoscopy; the bristol stool form scale
MeSH Terms: interventions — Bisacodyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group1 (Experimental): Subjects whose bristol stool forms are type 1 or 2, will receive standard bowel prep (2L PEG-ELP) the same-day of procedure.
  Interventions: Drug: Standard Bowel Prep (2L PEG-ELP)
- group2 (Experimental): Subjects whose bristol stool forms are type 1 or 2, will be asked to take standard bowel prep (2L PEG-ELP) the same-day of procedure and 10mg bisacodyl the day before procedure. ( 2L PEG-ELP and 10mg bisacodyl )
  Interventions: Drug: 2L PEG-ELP and 10mg bisacodyl
- group3 (Active Comparator): Subjects whose bristol stool forms are type 3 to 7, will receive standard bowel prep (2L PEG-ELP) the same-day of procedure.
  Interventions: Drug: Standard Bowel Prep (2L PEG-ELP)

INTERVENTIONS:
Drug: Standard Bowel Prep (2L PEG-ELP) — Subjects whose bristol stool forms are type 1 or 2, will be asked to take standard bowel prep (2L PEG-ELP) the same-day of procedure.
  Arms: group1
Drug: 2L PEG-ELP and 10mg bisacodyl — Subjects whose bristol stool forms are type 1 or 2, will be asked to take standard bowel prep (2L PEG-ELP) the same-day of procedure and 10mg bisacodyl the day before procedure.
  Arms: group2
Drug: Standard Bowel Prep (2L PEG-ELP) — Subjects whose bristol stool forms are type 3 to 7, will be asked to take standard bowel prep (2L PEG-ELP) the same-day of procedure.
  Arms: group3

SUMMARY:
The Bristol stool form scale ( BSFS) based tailored bowel cleansing regimen might be helpful to improve bowel cleansing quality before colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy is the standard approach for evaluating the colon currently. Thorough bowel cleansing is critical for adequate visualization of colonic mucosa during colonoscopy. Inadequate bowel cleansing results in adverse consequences for the examination, including lower adenoma detection rates, longer procedural time, lower cecal intubation rates, shorter intervals between examinations and an estimated 12-22% increase in overall colonoscopy cost.Unfortunately, despite advances in bowel preparation methods, up to one-third of all colonoscopies are reported to have an inadequate bowel preparation.

The Bristol stool form scale ( BSFS) was developed in 1988 by O'Donnell LJD et al and was widely applied in both gastrointestinal study and clinical practice. BSFS divides human stool into 7 different styles according to its moisture content. In our clinical work, we find that it is prone to gain poor bowel cleansing quality in patients who pass type 1or 2 stool. Unfortunately, there is lacking of study on tailored bowel preparation according to Bristol stool form scale. Thus, we intend to develop an easy, practical, BSFS based tailored bowel cleansing regimen, in order to serve clinical work and research.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older,
* scheduled to undergo elective outpatient colonoscopy,
* and were able to provide informed consent.

Exclusion Criteria:

* history of colorectal surgery
* severe colonic stricture or obstructing tumour
* dysphagia
* compromised swallowing reflex or mental status
* significant gastroparesis or gastric outlet obstruction
* known or suspected bowel obstruction or perforation
* severe chronic renal failure (creatinine clearance<30 ml/min
* severe congestive heart failure (New York Heart Association class III or IV)
* uncontrolled hypertension (systolic blood pressure>170 mm Hg, diastolic blood pressure>100 mm Hg)
* inflammatory bowel disease or megacolon
* dehydration
* disturbance of electrolytes
* pregnancy or lactation
* haemodynamically unstable
* unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Difference of scores rating by Boston Bowel Preparation Scale among 3 groups. | 9 months
  This is an established rating scale to evaluate the quality of bowel prep. The ratings will be compared among the 3 groups.

SECONDARY OUTCOMES:
Rate of non-compliance with instructions among 3 groups. | 9 months
Willingness to repeat bowel preparation among 3 groups. | 9 months
Polyp detection rate among 3 groups. | 9 months
Caecal intubation rate among 3 groups. | 9 months
Withdrawal time among 3 groups. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: li yanqing, PhD,MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China